CLINICAL TRIAL: NCT05870540
Title: A Quadruple Masked, Dose-Finding Study to Evaluate the Efficacy and Safety of Intranasal BPL-003, With Open Label Extension, in Patients With Treatment-Resistant Depression
Brief Title: BPL-003 Efficacy and Safety in Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPL-003-201
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: CORE: Quadruple masking: participant, Investigator, therapist, outcomes assessor and Sponsor.
  OLE: Open Label Extension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Low dose (Experimental): Active placebo comparator
  Interventions: Drug: BPL-003
- Medium dose (Experimental)
  Interventions: Drug: BPL-003
- High dose (Experimental)
  Interventions: Drug: BPL-003
- Monophasic (Experimental)
  Interventions: Drug: BPL-003
- Biphasic (Experimental)
  Interventions: Drug: BPL-003

INTERVENTIONS:
Drug: BPL-003 — A single dose administered intranasally
  Arms: High dose; Low dose; Medium dose; Monophasic
Drug: BPL-003 — A single dose administered intranasally (administered as 2 nasal sprays minutes apart)
  Arms: Biphasic

SUMMARY:
This is a Phase 2 study randomized, quadruple masked, multi-center study , with a Open Label Extension, designed to investigate the efficacy and safety of BPL-003 combined with psychological support in patients with treatment resistant depression (TRD).

DETAILED DESCRIPTION:
Approximately 200 eligible participants will receive a single dose of either low, medium, or high doses of BPL-003, given intranasally, with 8 weeks of follow up assessments. Following this participants may receive a second dose of either monophasic or biphasic dose of BPL-003, given intranasally, with another 8 weeks of follow up assessments.

Psychological support will be given before, during and after each dosing.

ELIGIBILITY:
Inclusion Criteria:

1. At least moderate major depressive disorder.
2. Diagnosed with TRD defined as failure to respond to an adequate dose and duration of at least 2 pharmacological treatments based on the MGH ATRQ assessment.
3. Hamilton Depression Rating Scale score ≥19 at Screening and Baseline.
4. CGI-S ≥4 at Screening and Baseline.
5. If currently taking antidepressant medications, willing and able to discontinue current antidepressants.

Exclusion Criteria:

1. Current or past history of schizophrenia, psychotic disorder including psychotic depression, bipolar disorder, delusional disorder, schizoaffective disorder, or any other severe psychiatric disorder.
2. Current personality disorders.
3. First-degree family history of schizophrenia, bipolar disorder, delusional disorder, or schizoaffective disorder.
4. Current alcohol or substance use disorder (other than caffeine or nicotine).
5. A participant who at any time has been unresponsive to ketamine, esketamine, an adequate course of treatment with electroconvulsive therapy, or has received vagal nerve stimulation or deep brain stimulation.
6. Suicidal ideation or behavior within the 12 months prior to the start of Screening or on Day 1 prior to dosing.
7. Suicide attempt and/or self-injurious behavior within the last 12 months prior to Screening.
8. Uncontrolled medical conditions e.g. hypo/hyperthyroidism, diabetes, renal failure.
9. History or current uncontrolled hypertension.
10. Seizure disorder or any seizure in the 2 years prior to Screening.
11. Has clinically significant results on ECG during the Screening.
12. Any nasal obstruction, blockage, or symptoms of congestion at the time of dosing that in the investigator's opinion may interfere with the administration of the study medication.
13. Female participants who are pregnant, lactating, or of childbearing potential and not willing to use adequate forms of contraception during the study.
14. Male participants who are sexually active and not willing to use adequate forms of contraception during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | 4 weeks
  High compared to low dose of BPL-003. The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. A higher MADRS score indicates more severe depression, and each item yields a score of 0-6.
OLE Primary Safety Outcome Measure | 8 weeks
  To determine the safety of a second dose of BPL-003 given with psychological support to participants with TRD as assessed by treatment-emergent adverse events.

SECONDARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | 1 week
  High compared to low dose of BPL-003. The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. A higher MADRS score indicates more severe depression, and each item yields a score of 0-6.
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | 4 weeks and 1 week
  Medium compared to low dose of BPL-003. The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. A higher MADRS score indicates more severe depression, and each item yields a score of 0-6.
Safety of BPL-003 given with psychological support as assessed by number and percentage of participants with adverse events | 8 weeks
Safety of BPL-003 given with psychological support as assessed by percentage of participants with clinically significant abnormal laboratory tests | 8 weeks
Safety of BPL-003 given with psychological support as assessed by percentage of participants with clinically significant abnormal vital sign measurements | 8 weeks
Safety of BPL-003 given with psychological support as assessed by percentage of participants with clinically significant ECG parameters compared | 8 weeks
Safety of BPL-003 given with psychological support as assessed by incidence of suicidal ideation or behavior | 8 weeks
Plasma levels of 5-MeO-DMT and its metabolites | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: VP & Head of Clinical Development, Study Director — Beckley Psytech Ltd
Locations (42):
- United States (19):
  - UAB School of Public Health, Department of Health Behavior, Birmingham, Alabama
  - Woodland Research Northwest, Rogers, Arkansas
  - Kadima Neuropsychiatry Institute, San Diego, California
  - San Francisco Insight and Integration Center, San Francisco, California
  - Pacific Neuroscience Institute, Treatment and Research in Psychedelics (TRIP) Program, Santa Monica, California
  - Wholeness Center, Fort Collins, Colorado
  - Segal Trials Center for Psychedelic and Cannabis Research, Lauderhill, Florida
  - Emory University, Brain Health Center, Department of Psychiatry and Behavioral Sciences, Atlanta, Georgia
  - CenExel ACMR, Atlanta, Georgia
  - CenExel iResearch, Decatur, Georgia
  - Sunstone Medical PC (Sunstone Therapies / Aquilino Cancer Center), Rockville, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - CenExel HRI, Berlin, New Jersey
  - New York State Psychiatric Institute, New York, New York
  - Portland Psychotherapy, Portland, Oregon
  - Insite clinical research, DeSoto, Texas
  - AIM Trials, Plano, Texas
  - Cedar Clinical Research, Draper, Utah
  - University of Wisconsin, Dept of Family Medicine & Community Health, Madison, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Dept. of Psychiatry and School Psychological Sciences, Monash University, Clayton, Victoria
  - NeuroCentrix Research, Melbourne
  - Royal Melbourne Hospital, University of Melbourne, Parkville
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - OVID Clinic, Augmented Psychotherapy, Berlin
  - Department of Psychiatry, University Hospital Frankfurt, Frankfurt am Main
  - Central Institute of Mental Health, Dept. of Molecular Neuroimaging, Mannheim
  - Universitätsklinik für Psychiatrie und Psychotherapie, Calwerstr. 14, Tübingen
- Poland (5):
  - Department of Psychiatry, UCK, Gdansk
  - Centrum Badań Klinicznych PI-House sp. z o.o., Gdansk
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Klinika Inventiva, Tuszyn
  - Department of Pharmacology and Physiology of CNS, Warsaw
- Spain (6):
  - Hospital del Mar, Barcelona
  - Parc Sanitari Sant Joan de Deu HD Numancia, Barcelona
  - Hospital Clinic de Barcelona, Psychiatry and Psychology Dept., Barcelona
  - Fundación de Investigación HM Hospital, Madrid
  - Centro de Salud Mental La Corredoria, Oviedo
  - Centro Salud San Juan, Salamanca
- United Kingdom (3):
  - NIHR Exeter Clinical Research Facility, Exeter
  - King's College London - Institute of Psychiatry, Psychology & Neuroscience (IoPPN) - Centre for Affective Disorders (CfAD), London
  - Clerkenwell Health, London

IPD SHARING:
Plan to Share IPD: No
Due to the GDPR, individual participant data will not be shared publicly. Group data will be presented in publication after study completion